CLINICAL TRIAL: NCT01734161
Title: A Prospective, Randomized, Double-Blinded Study to Evaluate the Efficacy of Intravenous Dexamethasone for Nausea Prophylaxis Prior to Duramorph and Bupivacaine Spinal Anesthesia for Scheduled Cesarean Section
Brief Title: Dexamethasone for the Prevention of Post-operative Nausea and Vomiting in Patients Undergoing Cesarean Sections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1207012632
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: cesarean section; nausea; vomiting; dexamethasone; postoperative nausea and vomiting; antiemetics
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): One dose of 8 mg of intravenous dexamethasone diluted in 50 ml of normal saline given as an infusion over 10 minutes.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): One dose of 50 ml of 0.9% normal saline that will be given as an infusion over 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 8mg IV dexamethesone given
  Other Names: Decadron
  Arms: Dexamethasone
Drug: Placebo — Subjects randomized to placebo receive 50cc normal saline
  Other Names: 50 ml 0.9% saline
  Arms: Placebo

SUMMARY:
Patients who present for scheduled (non-emergent) cesarean section will be given either intravenous dexamethasone or placebo prior to receiving a duramorph containing spinal anesthetic. The investigators will then compare the incidence of nausea and vomiting and the use of rescue anti-nausea medications in both groups. Our hypothesis is that patients receiving dexamethasone prior to duramorph containing spinal anesthesia for cesarean section will have a significantly lower incidence and severity of PONV at 0, 1, 3, 6, and 24 hours following surgery.

DETAILED DESCRIPTION:
Women having cesarean sections commonly experience post-operative nausea and vomiting (PONV). This can be partly attributed to the long acting morphine (duramorph) given in the anesthetic (either through the epidural or in the spinal anesthetic). Intravenous dexamethasone is a widely used steroid medication with a well-established safety profile which is the standard of care for the prevention of PONV for general anesthesia in both adult and pediatric surgical patients. Many studies have shown that when intravenous dexamethasone is administered before duramorph in the epidural, the incidence of nausea and vomiting following cesarean section is significantly reduced. However, when patients receive intravenous dexamethasone after duramorph in a spinal anesthetic, it does not reduce the incidence of nausea and vomiting. There are not any published studies where dexamethasone was administered before a spinal anesthetic. The investigators believe that if dexamethasone is given intravenously before duramorph in a spinal anesthetic it may reduce the incidence of nausea and vomiting. Patients who present for scheduled (non-emergent) cesarean section will be given either intravenous dexamethasone or placebo prior to receiving a duramorph containing spinal anesthetic. The investigators will then compare the incidence of nausea and vomiting and the use of rescue anti-nausea medications in both groups. Our hypothesis is that patients receiving dexamethasone prior to duramorph containing spinal anesthesia for cesarean section will have a significantly lower incidence and severity of PONV at 0, 1, 3, 6, and 24 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-46 presenting for scheduled primary or repeat cesarean sections and have consented to study

Exclusion Criteria:

* allergy to dexamethasone or morphine
* history of gastrointestinal disease
* history of severe nausea during pregnancy (hyperemesis gravidarum)
* use of anti-emetic in the past 24 hours
* history of gestational diabetes or diabetes mellitus
* history of hypertension prior to or during pregnancy
* presence of non-viable fetus

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kjaer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Allen TK, Jones CA, Habib AS. Dexamethasone for the prophylaxis of postoperative nausea and vomiting associated with neuraxial morphine administration: a systematic review and meta-analysis. Anesth Analg. 2012 Apr;114(4):813-22. doi: 10.1213/ANE.0b013e318247f628. Epub 2012 Feb 17. PMID 22344239
- [Background] Cardoso MM, Leite AO, Santos EA, Gozzani JL, Mathias LA. Effect of dexamethasone on prevention of postoperative nausea, vomiting and pain after caesarean section: a randomised, placebo-controlled, double-blind trial. Eur J Anaesthesiol. 2013 Mar;30(3):102-5. doi: 10.1097/EJA.0b013e328356676b. PMID 23022704
- [Background] Hamzei A, Basiri-Moghadam M, Pasban-Noghabi S. Effect of dexamethasone on incidence of headache after spinal anesthesia in cesarean section. A single blind randomized controlled trial. Saudi Med J. 2012 Sep;33(9):948-53. PMID 22964805
- [Derived] Selzer A, Pryor KO, Tangel V, O'Connell K, Kjaer K. The effect of intravenous dexamethasone on postoperative nausea and vomiting after Cesarean delivery with intrathecal morphine: a randomized-controlled trial. Can J Anaesth. 2020 Jul;67(7):817-826. doi: 10.1007/s12630-020-01582-y. Epub 2020 Jan 27. PMID 31989472
- See also: Nausea and Vomiting — http://www.nlm.nih.gov/medlineplus/nauseaandvomiting.html
- See also: Drug information for Dexamethasone — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0000050022&QV1=DEXAMETHASONE

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 61 | 61
Completed | 55 | 53
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 55 | 53 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (5.2) | 35.7 (3.7) | 35.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 108
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-operative Nausea and/or Vomiting
Description: The patient's self report of nausea and incidence of vomiting will be recorded intra-operatively, upon arrival to the PACU and at 1, 3, 6, 24, and 48 hours after surgery
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 55 | 53
Participants | 29 | 24

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/53
Other Adverse Events (participants affected / at risk) | 7/55 | 3/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=55) | Placebo (N=53)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) — Hypertension
incision site bleeding (Surgical and medical procedures) | 1 (1) | 0 — incision site bleeding
low body temperature (General disorders) | 2 (2) | 0 — low body temperature
post-op shivering (General disorders) | 1 (1) | 0 — post-op shivering
Tachycardia (Cardiac disorders) | 1 (1) | 0 — Tachycardia
Transfusion Required (Vascular disorders) | 1 (1) | 0 — Transfusion Required

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes